CLINICAL TRIAL: NCT03410121
Title: Phase IV Study Comparing Humeral or Thoracic Implantation of an Central Veinous Access by an Implantable Venous Access Device in Patients With Solid Tumors Requiring Intravenous Chemotherapy
Brief Title: Comparison of Humeral or Thoracic Implantation of an Central Veinous Access by an Implantable Venous Access Device in Patients With Solid Tumors Requiring Chemotherapy
Acronym: PACPAC-EPOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2016-4-46-002
Record Dates: First submitted 2018-01-18; First posted 2018-01-25 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor, Adult; Chemotherapy Treatment; Advanced or Metastasis Stage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard 1 : Thoracic location (Other): The intervention is characterized by the randomization into thoracic arm which means that patients will have an implantable Venous Access Device implanted into thoracic location
  Interventions: Device: IPolysite ® Mini série 3108 or Polysite ® Standard, série 4108.
- Standard 2 : Humeral location (Other): The intervention is characterized by the randomization into humeral arm which means that patients will have an implantable Venous Access Device implanted into humeral location
  Interventions: Device: Vital Port®Minititanium

INTERVENTIONS:
Device: IPolysite ® Mini série 3108 or Polysite ® Standard, série 4108. — Implantation of intravenous medical device in thoracic location
  Arms: Standard 1 : Thoracic location
Device: Vital Port®Minititanium — Implantation of intravenous medical device in humeral location
  Arms: Standard 2 : Humeral location

SUMMARY:
The aim of this study is to compare the humeral and thoracic implantation of a central venous access by an implantable device in patients with solids tumors who require intravenous chemotherapy. This is a monocentric randomized study. 572 patients will be recruited for 2 years. They will be randomized either in the thoracic implantation, either in the humeral implantation Due to the 1:3 randomization, 143 patients will be randomized in the humeral arm and 429 into the thoracic one. Number of complications related to the implantable device, medico-economic analysis as well as patient satisfaction will be assessed.

Every patients with solid tumor requiring medical device implantation for intravenous chemotherapy treatment will be eligible.

Both humeral and thoracic implantation of medical device are standard procedures. The randomization in a specific arm is the study procedure and is considered as an interventional study in France.

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid tumors at an Advanced or metastasis stage requiring placement of implantable catheter for intravenous chemotherapy treatment
* Older than 18 years
* Express signed consent

Exclusion Criteria:

* Life expectancy less than 12 months assessed by investigator
* Infection or uncontrolled suspected infection
* Medical contraindication to port implantation by catheter in thoracic or humeral location
* Pregnant or lactating women
* Abnormal coagulation
* Immunosuppressed patients (for example known hepatitis B or C, or known positive Human Immunodeficiency Virus due to the spreading risk)
* Patient not affiliated to the French social security
* Access time to the humeral or thoracic port placement higher than 15 days (from the randomization theoretical date)
* Protected Adult or adult deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2024-09-17 (Actual)

PRIMARY OUTCOMES:
Number of complications related to Implantable Venous Access Device | 3 months after medical device placement
  Number of complications that will be recorded by medical oncologist

CONTACTS AND LOCATIONS:
Overall Officials: Laurence CROUZET, MD, Principal Investigator — Centre Eugène Marquis, Rennes, France
Locations (1):
- Center Eugene Marquis, Rennes, Brittany Region, France

IPD SHARING:
Plan to Share IPD: No